CLINICAL TRIAL: NCT02583230
Title: Mobile Technology to Engage and Link Patients and Providers in Antidepressant Treatment (MedLink)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R34MH095907-FTML; R34MH095907 (NIH)
Record Dates: First submitted 2015-10-18; First posted 2015-10-22 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Antidepressant Medication; Adherence; Mobile Smartphone Intervention; Telemedicine; Primary Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MedLink (Experimental): For 8 weeks, the patient who is newly prescribed antidepressant medication will receive a mobile phone app (and a phone if they do not have a compatible Android phone) and a GSM enable pill bottle in order to provide and receive feedback regarding medication adherence.
  Interventions: Behavioral: MedLink System

INTERVENTIONS:
Behavioral: MedLink System — Patient adherence to anti depressant medication will be accomplished by 1) monitoring adherence and providing feedback to patient (e.g. prompting patient to take medication); 2) monitoring side effects and treatment response and providing in-the-moment feedback and support; 3) activating the patient to take appropriate action (e.g. call the prescribing physician) based upon monitoring data; 4) providing standardized education and positive reinforcement to the patient.
  The care team will be supported and activated by being provided 1) suggested guideline-congruent actions and 2) timely information regarding the patient's status.

SUMMARY:
The goal of this project is to develop and pilot a mobile smartphone delivered intervention that will improve antidepressant medication care by providing medication adherence monitoring and support to the patient, feedback on patient adherence and response to treatment to the primary care team, and information to both patients and providers on guideline-congruent care personalized to the patient's response to antidepressant medication.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is common and imposes a very high societal burden in terms of cost, morbidity, suffering, and mortality. While primary care is the de facto site for treatment of MDD, outcomes in primary care are poor. Two principal reasons for the poor outcomes in primary care are poor patient adherence to antidepressant medications (ADMs) and the failure of physicians to provide guideline-congruent care. This problem is aggravated by a lack of communication between patients and the care team.

A growing body of research indicates that primary care-centered strategies aimed at enhancing guideline-congruent care have not been effective. Interventions aimed at improving adherence in the patient have been successful in changing patient adherence behavior; however these frequently fail to improve depression outcomes, particularly when there is no intervention on the physician side to encourage optimization of ADMs. Recent developments in information and communications technologies (ICT) have opened new opportunities to improve health and mental health care, and to link patients and their providers. This study harnesses these advances to develop and pilot a system where ADM adherence will be passively measured using an electronic pill dispenser. The dispenser is connected to a mobile smartphone via Global System for Mobile Communications (GSM), so that targeted, timely reminders can be provided when the patient fails to take the ADM. When the patient is adherent, the patient will not be bothered with reminders. Depressive symptoms and side-effects will be periodically monitored weekly via the phone. Every 4 weeks, or if indicated (e.g intolerable side effects or urgent situations), primary care teams will receive notifications via the electronic medical record that include a summary of patient data on treatment response and side effects, guideline-congruent treatment recommendations based on patient data and a recommendation to contact the patient, if indicated. Simultaneously, a similar message will be provided to the patient, including feedback, possible treatment options, and a recommendation to contact the physician's office. Thus, both the patient and care team will be activated to provide, request and adhere to guideline-congruent care.

The aim of this 8 week field trial is to develop and pilot the MedLink system. Development will employ an iterative user-centered approach. Primary outcome will be patient adherence; secondary outcomes will be depression, system use, and usability and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Has been prescribed an antidepressant medication by a Primary Care Provider, but has not yet initiated treatment
* Has depression determined by primary care physician
* Is familiar with the use of mobile phones
* Is able and willing to carry the mobile phone
* Is able to speak and read English
* Is at least 18 years of age

Exclusion Criteria:

* Is current taking an antidepressant medication or has taken one in the previous 3 months
* Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of mobile phone
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance dependence, or other diagnosis for which participation in this trial is either inappropriate or dangerous. Patients with substance dependence diagnoses who have been clean and sober for 12 months will be admitted if otherwise eligible
* Is severely suicidal (has ideation, plan, and intent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University

RESULTS

PARTICIPANT FLOW:
Groups:
- MedLink: For 8 weeks, the patient who is newly prescribed antidepressant medication will receive a mobile phone app (and a phone if they do not have a compatible Android phone) and a GSM enabled pill bottle in order to provide and receive feedback regarding medication adherence.
  MedLink System: Patient adherence to anti depressant medication will be accomplished by 1) monitoring adherence and providing feedback to patient (e.g. prompting patient to take medication); 2) monitoring side effects and treatment response and providing in-the-moment feedback and support; 3) activating the patient to take appropriate action (e.g. call the prescribing physician) based upon monitoring data; 4) providing standardized education and positive reinforcement to the patient.
  The care team will be supported and activated by being provided 1) suggested guideline-congruent actions and 2) timely information regarding the patient's status.
Period: Overall Study
Arm/Group | MedLink
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for enrolled participants.
Arm/Group | MedLink
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 7
  Living with significant other | 1
  Married/Domestic partner | 3
Education [Count of Participants; unit: Participants]
  Some high school | 1
  Completed high school | 1
  4-year college (BA, BS) | 5
  Master's degree | 4
Employment status [Count of Participants; unit: Participants]
  Employed | 7
  Unemployed | 1
  Retired | 2
  Student | 1
Mobile device [Count of Participants; unit: Participants]
  Personal device | 4
  Study provided device | 7

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Antidepressant Medication
Description: Number of days medication was taken when a dose was expected. Measured through % of days adherent on Wisepill pillbox as well as 2. Self-reported adherence: Patient Adherence Questionnaire (PAQ).
Time Frame: 8 weeks
Measure: Number; unit: % of days adherent
Arm/Group | MedLink
Number analyzed (Participants) | 11
% of days adherent | 82.0

2. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome. Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MedLink
Number analyzed (Participants) | 11
units on a scale
  Baseline | 12.0 (4.0)
  Week 4 | 5.3 (4.6)
  Week 8 | 3.5 (6.5)
Statistical Analysis 1: Comparison: MedLink; Test type: Superiority; p = .0005, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel test was used to evaluate the change in PHQ-9 total scores over the eight-week study period

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology Clinician Rating (QIDS-C)
Description: This measure assesses depressive symptom severity. The total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV MDD (major depressive disorder) criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes (Rush et al. 2003). Sixteen items are used to rate the nine criterion symptom domains of a major depressive episode. Each item is rated 0-3. For symptom domains that require more than one item, the highest score of the item relevant for each domain is taken. The total score ranges from 0-27. Higher values represent a worse outcome. Specifically, scores of 0-5 indicate no depression; 6-10 is mild; 11-15 is moderate; 16-20 is severe; and 21-27 is very severe.
Time Frame: Baseline, Week 4, and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MedLink
Number analyzed (Participants) | 11
units on a scale
  Baseline | 11.6 (3.7)
  Week 4 | 7.6 (5.6)
  Week 8 | 4.6 (4.0)
Statistical Analysis 1: Comparison: MedLink; Test type: Superiority; p = .0008, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel test was used to evaluate the change in QIDS total scores over the eight-week study period

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- MedLink: For 8 weeks, the patient who is newly prescribed antidepressant medication will receive a mobile phone app (and a phone if they do not have a compatible Android phone) and a GSM enable pill bottle in order to provide and receive feedback regarding medication adherence.
  MedLink System: Patient adherence to anti depressant medication will be accomplished by 1) monitoring adherence and providing feedback to patient (e.g. prompting patient to take medication); 2) monitoring side effects and treatment response and providing in-the-moment feedback and support; 3) activating the patient to take appropriate action (e.g. call the prescribing physician) based upon monitoring data; 4) providing standardized education and positive reinforcement to the patient.
  The care team will be supported and activated by being provided 1) suggested guideline-congruent actions and 2) timely information regarding the patient's status.
Arm/Group | MedLink
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes